CLINICAL TRIAL: NCT00000603
Title: Cord Blood Stem Cell Transplantation Study (COBLT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Purpose: Treatment
Other Study IDs: 316
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2008-01

CONDITIONS: Anemia, Aplastic; Fanconi Anemia; Hematologic Diseases; Leukemia; Neoplasms; Severe Combined Immunodeficiency; Hematopoietic Stem Cell Transplantation; Myelodysplastic Syndromes
MeSH Terms: conditions — Anemia, Aplastic; Fanconi Anemia; Hematologic Diseases; Leukemia; Neoplasms; Severe Combined Immunodeficiency; Myelodysplastic Syndromes | interventions — Stem Cell Transplantation

INTERVENTIONS:
Procedure: stem cell transplantation

SUMMARY:
To evaluate if HLA-mismatched, unrelated-donor umbilical cord blood stem and progenitor cell units (UCBU) offered a clinically acceptable alternative to matched unrelated-donor allogeneic bone marrow for transplantation with 180-day disease free survival as the endpoint. HLA typing was performed using DNA-base high resolution methods to determine HLA alleles. Patients with "true" HLA 3/6 and 4/6 matches were evaluated. In addition, a separate study in adults addressed the problem of limited cell dose and engraftment failure. The study was not planned as a randomized comparative clinical trial. Instead, it is a phase II/III efficacy study.

DETAILED DESCRIPTION:
BACKGROUND:

Bone marrow transplantation is an effective therapy for a variety of genetic and hematologic disorders. Donated bone marrow, which provides a source of stem and progenitor cells for bone marrow reconstitution, is obtained either from related donors, usually HLA-matched siblings, or from HLA-matched unrelated donors. Because of the limited availability of HLA-matched related donors, HLA-matched unrelated donors are frequently the only alternative source of bone marrow for transplantation. To provide matched volunteer bone marrow donors for unrelated recipients, the National Marrow Donor Program (NMDP) was established in 1986 to develop a national Registry of HLA-typed individuals who agree to donate bone marrow if needed. More than 3 million potential marrow donors are now enrolled. A limitation of the registry approach is the time needed to identify a donor and complete the necessary clinical evaluation and laboratory testing for histocompatibility, infectious diseases, and general good health. Moreover, a certain proportion of potential donors change their minds or otherwise become unavailable between the time they enter the Registry and the time they are called as a preliminary match for a patient. Another disadvantage is the marrow harvesting procedure which requires the normal donor to be hospitalized and given general anesthesia in an operating room. Finally, the NMDP Registry consists of potential donors that are primarily of European Caucasian ancestry. Although great strides have been made in increasing the numbers of African-Americans, Hispanics, Asian-Americans, and Native Americans, it is still more difficult to find matches for these ethnic minorities than for Caucasian patients.

Human umbilical cord blood is an alternative source of hematopoietic stem and progenitor cells capable of reconstituting the bone marrow of recipients with a variety of diseases. Cord blood stem and progenitor cells from related donors have been successfully transplanted world-wide in children with genetic or hematologic diseases. These results suggested that cord blood from unrelated, HLA-matched donors also can be used for patients who need a transplant but don't have a related donor. The existing problems in unrelated-donor bone marrow transplantation with donor recruitment, bone marrow harvesting, and matching for antigens peculiar to a particular ethnic group would be reduced if typed, tested, and frozen umbilical cord blood could be made easily and rapidly available. Such a system, which could complement or partially replace the present process, has been shown to be feasible. In an NHLBI-sponsored program, investigators have collected and cryopreserved a bank of about 9,000 human UCBUs. In addition, successful searches and matches (including many 4/6 antigen matches) have resulted in more than 900 unrelated-donor, UCBU transplants to date. Preliminary data from both these unrelated-donor and other related-donor cord blood transplants suggest that there is less GvHD than if the source of the graft were adult bone marrow. The severity of GvHD also seems less even in highly mismatched recipients. One important question is whether or not 3/6 HLA matched transplants in children will have acceptable 180-day disease free survival. It also remains to be determined if the graft-vs-leukemia effect is also less or if unrelated-donor cord blood grafts are as durable as those from matched, related-donors. Most transplants conducted thus far have been in children. Hence another important question is whether or not there are sufficient numbers of stem cells in cord blood to support transplantation to an unrelated adult.

The initiative was proposed by the Division of Blood Diseases and Resources staff and approved by the February 1995 National Heart, Lung, and Blood Advisory Council. The Requests for Proposals were released in June 1995. Contracts were awarded September 30, 1997.

DESIGN NARRATIVE:

The study is multicenter, with six Cord Blood Transplant Centers (CBTCs), two collecting and storage centers (Cord Blood Banks -- CBBs) and one Coordinating Center. Each CBB used the same protocol for recruiting donors, collecting, processing, testing, storage, retrieval from storage, reprocessing from the frozen state, and shipping. Each participating CBTC used the same patient selection criteria, preparative regimen for patients in the same class, initial graft-versus-host disease (GvHD) prophylaxis, indications for the use of cytokines, definitions for events and complications, and methods for evaluating immune reconstitution. The main study evaluated the impact of HLA 3/6 and 4/6 matching on outcome. The primary endpoint was 180-day disease free survival after UCBU transplantation. Secondary endpoints included engraftment, the frequency and severity of acute and chronic GvHD with stratification by degree of HLA match, overall survival, and immunologic reconstitution. Data were collected on banked UCBUs to define unit quality by nucleated cell count and flow cytometry of surface markers to identify effects on patient outcome. Recruitment ended December 31, 2003 with the accrual of 326 subjects. .

ELIGIBILITY:
Mothers of Infant-donors must complete a medical history form, have an uncomplicated delivery, and deliver at UCLA or Duke.

Patients are those who need a transplant but don't have a matched marrow donor or can't wait to find one.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1996-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelly Carter — The Emmes Company, LLC; Joanne Kurtzberg — Duke University

REFERENCES:
- [Background] Wagner JE, Kurtzberg J. Banking and transplantation of unrelated donor umbilical cord blood: status of the National Heart, Lung, and Blood Institute-sponsored trial. Transfusion. 1998 Sep;38(9):807-9. doi: 10.1046/j.1537-2995.1998.38998408998.x. No abstract available. PMID 9738618
- [Background] Fraser JK, Cairo MS, Wagner EL, McCurdy PR, Baxter-Lowe LA, Carter SL, Kernan NA, Lill MC, Slone V, Wagner JE, Wallas CH, Kurtzberg J. Cord Blood Transplantation Study (COBLT): cord blood bank standard operating procedures. J Hematother. 1998 Dec;7(6):521-61. doi: 10.1089/scd.1.1998.7.521. PMID 9919946
- [Background] Laughlin MJ, Barker J, Bambach B, Koc ON, Rizzieri DA, Wagner JE, Gerson SL, Lazarus HM, Cairo M, Stevens CE, Rubinstein P, Kurtzberg J. Hematopoietic engraftment and survival in adult recipients of umbilical-cord blood from unrelated donors. N Engl J Med. 2001 Jun 14;344(24):1815-22. doi: 10.1056/NEJM200106143442402. PMID 11407342
- [Background] Barker JN, Wagner JE. Umbilical cord blood transplantation: current practice and future innovations. Crit Rev Oncol Hematol. 2003 Oct;48(1):35-43. doi: 10.1016/s1040-8428(03)00092-1. PMID 14585482
- [Background] Staba SL, Escolar ML, Poe M, Kim Y, Martin PL, Szabolcs P, Allison-Thacker J, Wood S, Wenger DA, Rubinstein P, Hopwood JJ, Krivit W, Kurtzberg J. Cord-blood transplants from unrelated donors in patients with Hurler's syndrome. N Engl J Med. 2004 May 6;350(19):1960-9. doi: 10.1056/NEJMoa032613. PMID 15128896
- [Background] Laughlin MJ, Eapen M, Rubinstein P, Wagner JE, Zhang MJ, Champlin RE, Stevens C, Barker JN, Gale RP, Lazarus HM, Marks DI, van Rood JJ, Scaradavou A, Horowitz MM. Outcomes after transplantation of cord blood or bone marrow from unrelated donors in adults with leukemia. N Engl J Med. 2004 Nov 25;351(22):2265-75. doi: 10.1056/NEJMoa041276. PMID 15564543
- [Background] Cornetta K, Laughlin M, Carter S, Wall D, Weinthal J, Delaney C, Wagner J, Sweetman R, McCarthy P, Chao N. Umbilical cord blood transplantation in adults: results of the prospective Cord Blood Transplantation (COBLT). Biol Blood Marrow Transplant. 2005 Feb;11(2):149-60. doi: 10.1016/j.bbmt.2004.11.020. PMID 15682076
- [Background] Wall DA, Carter SL, Kernan NA, Kapoor N, Kamani NR, Brochstein JA, Frangoul H, Goyal RK, Horan JT, Pietryga D, Wagner JE, Kurtzberg J; COBLT Steering Committee. Busulfan/melphalan/antithymocyte globulin followed by unrelated donor cord blood transplantation for treatment of infant leukemia and leukemia in young children: the Cord Blood Transplantation study (COBLT) experience. Biol Blood Marrow Transplant. 2005 Aug;11(8):637-46. doi: 10.1016/j.bbmt.2005.05.003. PMID 16041314
- [Background] Cairo MS, Wagner EL, Fraser J, Cohen G, van de Ven C, Carter SL, Kernan NA, Kurtzberg J. Characterization of banked umbilical cord blood hematopoietic progenitor cells and lymphocyte subsets and correlation with ethnicity, birth weight, sex, and type of delivery: a Cord Blood Transplantation (COBLT) Study report. Transfusion. 2005 Jun;45(6):856-66. doi: 10.1111/j.1537-2995.2005.04429.x. PMID 15934982
- [Background] Kurtzberg J, Cairo MS, Fraser JK, Baxter-Lowe L, Cohen G, Carter SL, Kernan NA. Results of the cord blood transplantation (COBLT) study unrelated donor banking program. Transfusion. 2005 Jun;45(6):842-55. doi: 10.1111/j.1537-2995.2005.04428.x. PMID 15934981
- [Derived] Kurtzberg J, Prasad VK, Carter SL, Wagner JE, Baxter-Lowe LA, Wall D, Kapoor N, Guinan EC, Feig SA, Wagner EL, Kernan NA; COBLT Steering Committee. Results of the Cord Blood Transplantation Study (COBLT): clinical outcomes of unrelated donor umbilical cord blood transplantation in pediatric patients with hematologic malignancies. Blood. 2008 Nov 15;112(10):4318-27. doi: 10.1182/blood-2007-06-098020. Epub 2008 Aug 21. PMID 18723429
- Available data/document: Individual Participant Data Set: COBLT — http://biolincc.nhlbi.nih.gov/studies/coblt/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/coblt/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/coblt/
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/coblt/